CLINICAL TRIAL: NCT00656201
Title: Comparison of Crinone 8% Intravaginal Gel or Intramuscular Progesterone Supplementation for In Vitro Fertilization (IVF) and Embryo Transfer (ET) Cycles in Women Under Age 40 Years Old
Brief Title: Comparison of Crinone 8% Intravaginal Gel and IM Progesterone Supplementation for In Vitro Fertilization (IVF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Elena Hesina Yanushpolsky, MD, Assistant Professor of Ob/Gyn, BWH and Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWH 2003p000075
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2011-09-20 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Infertility
Keywords: Infertility; In vitro fertilization; Embryo transfer; Crinone; Intramuscular Progesterone; Progesterone support
MeSH Terms: conditions — Infertility | interventions — Crinone; Vaginal Creams, Foams, and Jellies; Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crinone 8% Vaginal Gel (Active Comparator): Crinone 8% (90 mg of micronized progesterone in a bioadhesive vaginal gel contained in a single use, one piece applicator) once a day beginning the second day following oocyte retrieval (Study Group A) continuing until the pregnancy test is negative or until the 10th week of pregnancy.
  Interventions: Drug: Crinone 8% Vaginal Gel
- Intramuscular Progesterone (Active Comparator): Progesterone-50 mg intramuscularly once a day beginning the day after oocyte retrieval continuing until the pregnancy test is negative or if positive, switching to Crinone 8% intravaginal gel until the 10th week of pregnancy.
  .
  Interventions: Drug: Intramuscular Progesterone

INTERVENTIONS:
Drug: Crinone 8% Vaginal Gel — Crinone 8% (90 mg of micronized progesterone in a bioadhesive vaginal gel contained in a single use, one piece applicator) once a day beginning the second day following oocyte retrieval (Study Group A) continuing until the pregnancy test is negative or until the 10th week of pregnancy.
  Other Names: IVF-ET; Pregnancy; luteal phase support; Crinone; Intramuscular progesterone; vaginal progesterone
  Arms: Crinone 8% Vaginal Gel
Drug: Intramuscular Progesterone — Progesterone-50 mg intramuscularly once a day beginning the day after oocyte retrieval continuing until the pregnancy test is negative or if positive, switching to Crinone 8% intravaginal gel until the 10th week of pregnancy.
  Other Names: Other Names:; IVF-ET; Pregnancy; luteal phase support; Crinone; vaginal progesterone
  Arms: Intramuscular Progesterone

SUMMARY:
The goal of this research study is to compare the pregnancy rates for two different types of progesterone supplementation after in-vitro fertilization (IVF).

DETAILED DESCRIPTION:
The aim is to test the hypothesis that the pregnancy rates of women under age 40 undergoing an in vitro fertilization and embryo transfer (IVF-ET) cycle are not different with respect to the administration of progesterone (Crinone 8%, intravaginal gel versus intramuscular progesterone).

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (21-39) with infertility who are appropriate candidates for IVF/ET and have an FSH < 15 mIU/ml
* Women 21 to 39 years of age who have been assigned to stimulation of 2 to 8 amps of Luteal Lupron/FSH or Luteal Lupron FSH/HMG.

Exclusion Criteria:

* Women who have had more than 3 previous IVF/ET cycles

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 468 (Actual)
Dates: Start 2003-07; Primary Completion 2008-11 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena H Yanushpolsky, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yanushpolsky E, Hurwitz S, Greenberg L, Racowsky C, Hornstein M. Crinone vaginal gel is equally effective and better tolerated than intramuscular progesterone for luteal phase support in in vitro fertilization-embryo transfer cycles: a prospective randomized study. Fertil Steril. 2010 Dec;94(7):2596-9. doi: 10.1016/j.fertnstert.2010.02.033. Epub 2010 Mar 27. PMID 20347079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients starting an IVF cycle will receive a letter from their physician and Dr. Yanushpolsky. We will include a copy of the consent form. This letter will briefly describe the study and will have an opt out paragraph. Patients fulfilling inc/exc criteria will be approached on the day of their oocyte retrieval by a study coordinator.
Pre-assignment Details: The participant may not qualify for enrollment if there were no eggs fertilized, or no embryos transfered, or all embryos frozen.
Period: Overall Study
Arm/Group | Crinone 8% Vaginal Gel | Intramuscular Progesterone
Started | 235 | 233
Completed | 206 | 201
Not Completed | 29 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crinone 8% Vaginal Gel | Intramuscular Progesterone | Total
Number analyzed (Participants) | 235 | 233 | 468
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 235 | 233 | 468
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.0 (3.3) | 34.2 (3.5) | 34.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235 | 233 | 468
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 235 | 233 | 468

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pregnant Patients After IVF Treatments
Description: Percentage of pregnant patients after IVF treatments who received either Crinone or IM Progesterone after oocyte retrieval
Time Frame: 16 weeks
Population: Number of participants for analysis was determined by completion of the IVF cycle using the specified medications, either Crinone or IM Progesterone
Measure: Number; unit: percentage of participants
Arm/Group | Crinone 8% Vaginal Gel | Intramuscular Progesterone
Number analyzed (Participants) | 206 | 201
percentage of participants | 66 [80 to 180] | 62 [80 to 180]
Statistical Analysis 1: Comparison: Crinone 8% Vaginal Gel vs Intramuscular Progesterone; Test type: Non-Inferiority or Equivalence — This was an equivalence comparison. The study was designed to detect a 14% pregnancy difference between the arms with 80% power and one interim analysis using O'Brien-Fleming parameters and an experiment-wise alpha level of 5%; p < 0.05, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.8 to 1.8] — Crinone is the numerator and IM Progesterone is the denominator

ADVERSE EVENTS:
Time Frame: From day of consent through 6 weeks of participation
Arm/Group | Crinone 8% Vaginal Gel | Intramuscular Progesterone
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/201
Other Adverse Events (participants affected / at risk) | 0/206 | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No